CLINICAL TRIAL: NCT00682786
Title: Genotype-directed Neoadjuvant Chemoradiation for Rectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-0561
Record Dates: First submitted 2008-04-11; First posted 2008-05-22 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Rectal Carcinoma
Keywords: rectal; rectum; cancer; carcinoma
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Carcinoma | interventions — Fluorouracil; Radiation; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) (Experimental): Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
  Interventions: Drug: 5FU; Radiation: Radiation; Procedure: Surgery of resectable lesions
- Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4) (Experimental): Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Irinotecan 50 mg/m2 IV weekly for 5 doses.
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
  Interventions: Drug: 5FU; Radiation: Radiation; Procedure: Surgery of resectable lesions; Drug: Irinotecan

INTERVENTIONS:
Drug: 5FU
  Other Names: Fluorouracil; 5-fluorouracil
Radiation: Radiation
Procedure: Surgery of resectable lesions
Drug: Irinotecan
  Other Names: Camptosar
  Arms: Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4)

SUMMARY:
Determine if genotype-directed neoadjuvant chemoradiation, using information from the thymidylate synthase promoter polymorphism, result in a greater degree of tumor downstaging in high risk patients compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum
* Lesion evaluated by surgeon and found to be resectable
* Stage T3 or T4 disease on radiography or ultrasound
* Karnofsky Performance Status at >60
* Laboratory criteria:

  * Absolute neutrophil count >= 1.5 K
  * Platelets >= 100 K
  * Total Bilirubin <= 2.0;
  * SGOT and Alkaline Phosphatase <= 2 x upper limit of normal
  * Creatinine < 2.0
* Informed consent signed
* Patients with distant metastatic disease will be eligible if they satisfy all other conditions.

Exclusion Criteria:

* Pregnant women, children < 18 years, or patients unable to give informed consent
* Patients with a past history of pelvic radiotherapy.
* Patients with prior malignancy in the past 5 years except: skin cancer or in-situ cervical cancer. However, patients with synchronous adenocarcinomas are eligible provided either (a) the synchronous adenocarcinoma was in a removed pedunculated polyp and did not invade the stalk or (b) the synchronous adenocarcinoma was in a removed polyp that lay within the surgical field (extent of resection would not be changed) or (c) the synchronous adenocarcinoma is smaller than the index rectal cancer and lies completely within the radiation field (clinically favorable second lesion and the extend of radiation and surgery would not be changed).
* Patients with known allergy to 5-fluorouracil or irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2002-10; Primary Completion 2008-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study opened on 10/07/2002 and the study closed to enrollment on 10/23/2008.
Period: Overall Study
Arm/Group | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4)
Started | 98 | 37
Completed | 96 | 34
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Did not receive irinotecan | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Good Risk (TYMS*2/*2, *2/*3, *2/*4): Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
- Poor Risk (TYMS*3/*3, *3/*4): Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Irinotecan 50 mg/m2 IV weekly for 5 doses.
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
- Total: Total of all reporting groups
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4) | Total
Number analyzed (Participants) | 98 | 37 | 135
Age, Continuous [Median (Full Range); unit: years] | 55 [32 to 85] | 59 [26 to 77] | 56 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 24 | 93
  Male | 29 | 13 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  White | 86 | 29 | 115
  African American | 10 | 8 | 18
  Hispanic | 1 | 0 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 98 | 37 | 135
Thymidylate Synthase Enhancer Region (TSER) genotype [Number; unit: participants]
  *2/*2 | 26 | 0 | 26
  *2/*3 | 71 | 0 | 71
  *2/*4 | 1 | 0 | 1
  *3/*3 | 0 | 35 | 35
  *3/*4 | 0 | 2 | 2
Performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Grade 0 Fully active able to carry on all predisease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (light house work/office work)
  2. Ambulatory, capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours
  3. Capable of limited selfcare, confined to bed/chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on selfcare. Totally confined to bed/chair
  5. Dead
  participants
    0 | 63 | 26 | 89
    1 | 34 | 11 | 45
    2 | 1 | 0 | 1
Baseline Stage [Number; unit: participants] — * T describes how far the primary tumor has grown into the wall of the intestine and whether it has grown into nearby areas.
  * N describes the extent of spread to nearby lymph nodes.
  * M indicates whether the cancer has spread to other organs of the body.
  Numbers or letters appear after T, N, and M to provide more details about each of these factors. The numbers 0 through 4 indicate increasing severity. The letter X means "cannot be assessed because the information is not available."
  participants
    Stage IIA (T3, N0, M0) | 24 | 10 | 34
    Stage IIB (T4, N0, M0) | 3 | 0 | 3
    Stage IIIA (T1-2, N1, M0) | 1 | 0 | 1
    Stage IIIB (T3-4, N1, M0) | 53 | 19 | 72
    Stage IIIC (T-any, N2, M0) | 3 | 3 | 6
    Stage IV (T-any, N-any, M1) | 14 | 5 | 19
Baseline clinical T stage [Number; unit: participants]
  T1-2 | 2 | 0 | 2
  T3 | 77 | 32 | 109
  T4 | 19 | 5 | 24
Baseline clinical N stage [Number; unit: participants]
  N0 | 30 | 11 | 41
  N1 | 64 | 22 | 86
  N2 | 4 | 4 | 8
Baseline clinical M stage [Number; unit: participants]
  M0 | 84 | 32 | 116
  M1 | 14 | 5 | 19
Clinical staging modality [Number; unit: participants]
  Endoscopic ultrasound | 60 | 21 | 81
  CT Scan +/- PET Scan | 22 | 6 | 28
  MRI | 16 | 10 | 26
Tumor distance from anal verge (cm) [Number; unit: participants]
  <5 | 33 | 12 | 45
  5-10 | 57 | 21 | 78
  >10 | 8 | 4 | 12
Tumor grade [Number; unit: participants]
  Well differentiated | 8 | 4 | 12
  Moderately differentiated | 68 | 25 | 93
  Poorly differentiated | 17 | 7 | 24
  Not reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Tumor Downstaging Compared With Historical Controls.
Description: Tumor downstaging (DS) is defined as a decrease in the T stage of the primary tumor by at least 1.
  Historical studies demonstrate a DS rate of 45%.
Time Frame: 1 year after enrollment
Population: 8 not evaluable in Good Risk arm-(1)death before surgery (1)clinical CR w/o surgery (1)refused surgery (2)not resectable (2)withdrew consent (1)delayed surgery and given FOLFOX
  6 not evaluable in Poor Risk arm-(1) death prior to surgery (1)clinical CR no surgery (1)refused surgery (2)withdrew consent (1)not given irinotecan by treating physician
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4)
Number analyzed (Participants) | 90 | 31
percentage of participants | 64.4 [54.1 to 74.6] | 64.5 [43.7 to 78.9]

2. Secondary Outcome: Complete Response Rates
Description: Complete tumor response is defined as the absence of any viable tumor in the rectum (ypT0).
  Pathologic complete response (pCR) is defined as the absence of any viable tumor in the rectum or in the perirectal lymph nodes (ypT0N0).
  pCR rate of historical controls is 8%-14%.
Time Frame: 1 year after enrollment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4)
Number analyzed (Participants) | 90 | 31
percentage of participants
  ypT0 | 20 | 41.9
  pCR | 18.9 | 35.5

3. Secondary Outcome: Define Patient Quality of Life Prior to and Following Neoadjuvant Chemoradiation.
Description: The questionnaire is encouraged but not required.
Time Frame: Prior to start of study treatment and 3-6 weeks post completion of radiation therapy
Population: The data was not collected for this outcome measure as the questionnaire was encouraged but not required.
Arm/Group | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Determine Patient Fears and Expectations of Pharmacogenetics.
Description: The questionnaire is encouraged but not required.
Time Frame: Prior to start of study treatment and 3-6 weeks post completion of radiation therapy
Population: The data was not collected for this outcome measure as the questionnaire was encouraged but not required.
Arm/Group | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4)
Number analyzed (Participants) | 0 | 0

5. Post Hoc Outcome: Toxicities by Genotype Group (Good Risk Versus Poor Risk)
Description: Grade 3 to 4 toxicities related to treatment and surgery using CTC Version 2.0.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: Two of the patients in the Good Risk arm withdrew consent and are not included. Two of the patients in the Poor Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4)
Number analyzed (Participants) | 96 | 35
participants
  Nausea | 0 | 1
  Vomiting | 0 | 1
  Diarrhea | 17 | 16
  Dehydration | 3 | 7
  Mucositis | 4 | 1
  GI bleed | 2 | 0
  Ileitis | 0 | 1
  Enteritis | 1 | 0
  Dyspnea | 1 | 0
  Neutropenia | 0 | 1
  Anemia | 3 | 3
  Pain | 3 | 4
  Perforation | 2 | 1
  Pelvic abscess | 0 | 2
  PPE | 0 | 1
  Crohn's flare | 1 | 0
  Syncope | 2 | 0
  Rash | 2 | 0
  Fatigue | 1 | 0
  Atrial fibrillation | 1 | 0
  Infection | 1 | 1
  Headache | 1 | 0
  Small bowel obstruction | 1 | 0

6. Post Hoc Outcome: Overall Survival
Description: Analyzed using Kaplan-Meier Models.
Time Frame: 1 year, 2 years, and 3 years
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4)
Number analyzed (Participants) | 96 | 35
percentage of participants
  1 year | 96.9 | 94.3
  2 years | 80.6 | 94.3
  3 years | 78.2 | 83.6

7. Post Hoc Outcome: Relapse-free Survival
Description: Analyzed using Kaplan-Meier Models.
Time Frame: 1 year, 2 years, and 3 years
Population: 14 patients in the Good Risk arm had metastatic rectal cancer at time of enrollment are not included in this analyses.
  3 patients in the Poor Risk arm had metastatic rectal disease before surgery and are included in this analyses.
  2 of the patients in the Good Risk arm and Poork Risk arm withdrew consent and are not included.
Measure: Number; unit: percentage of participants
Arm/Group | Good Risk (TYMS*2/*2, *2/*3, *2/*4) | Poor Risk (TYMS*3/*3, *3/*4)
Number analyzed (Participants) | 82 | 32
percentage of participants
  1 year | 85.2 | 87.0
  2 years | 78.3 | 80.5
  3 years | 73.4 | 72.4

8. Post Hoc Outcome: Associations Between MTHFR Genotypes and Grade 3-4 Diarrhea and/or Mucositis (Good Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
  MTHFR gene = methylenetetrahydrofolate reductase (NAD(P)H)
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Good Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Groups:
- Without Grade 3-4 Diarrhea and/or Mucositis; With Grade 3-4 Diarrhea and/or Mucositis: Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 75 | 21
participants
  CC (MTHFR 677C>T) | 34 | 5
  CT (MTHFR 677C>T) | 34 | 12
  TT (MTHFR 677C>T) | 7 | 4

9. Post Hoc Outcome: Associations Between MTHFR Genotypes and Grade 3-4 Diarrhea and/or Mucositis (Poor Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Poor Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Groups:
- Without Grade 3-4 Diarrhea and/or Mucositis; With Grade 3-4 Diarrhea and/or Mucositis: Radiation 45 Gy in 25 fractions to the pelvis.
  5FU CIVI 225 mg/m2/day by CIVI during radiation
  Irinotecan 50 mg/m2 IV weekly for 5 doses.
  Surgery 6-10 weeks after completion of preoperative radiation if disease has become resectable.
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 19 | 16
participants
  CC (MTHFR 677C>T) | 12 | 9
  CT (MTHFR 677C>T) | 6 | 7
  TT (MTHFR 677C>T) | 1 | 0

10. Post Hoc Outcome: Associations Between MTHFR Genotypes and Grade 3-4 Diarrhea and/or Mucositis (Good Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Good Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 75 | 21
participants
  AA (MTHFR 1298A>C) | 26 | 15
  AC (MTHFR 1298A>C) | 41 | 4
  CC (MTHFR 1298A>C) | 8 | 2

11. Post Hoc Outcome: Associations Between MTHFR Genotypes and Grade 3-4 Diarrhea and/or Mucositis (Poor Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Poor Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 19 | 16
participants
  AA (MTHFR 1298A>C) | 9 | 8
  AC (MTHFR 1298A>C) | 9 | 6
  CC (MTHFR 1298A>C) | 1 | 2

12. Post Hoc Outcome: Associations Between MTHFR Haplotypes and Grade 3-4 Diarrhea and/or Mucositis (Good Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Good Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 75 | 21
participants
  677C-1298A | 33 | 12
  677C-1298C | 49 | 6
  677T-1298A | 40 | 16

13. Post Hoc Outcome: Associations Between MTHFR Haplotypes and Grade 3-4 Diarrhea and/or Mucositis (Poor Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Poor Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 19 | 16
participants
  677C-1298A | 15 | 11
  677C-1298C | 10 | 8
  677T-1298A | 7 | 7

14. Post Hoc Outcome: Associations Between MTHFR Diplotypes and Grade 3-4 Diarrhea and/or Mucositis (Good Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Good Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 75 | 21
participants
  CA-CA | 13 | 2
  CA-CC | 14 | 1
  CA-TA | 6 | 9
  CC-CC | 7 | 2
  CC-TA | 27 | 3
  CC-TC | 1 | 0
  TA-TA | 7 | 4

15. Post Hoc Outcome: Associations Between MTHFR Diplotypes and Grade 3-4 Diarrhea and/or Mucositis (Poor Risk Group)
Description: Genomic DNA was isolated from whole blood using the Puregene DNA isolation kit.
Time Frame: First day of treatment through 30 days after completion of surgery
Population: 2 of the patients in the Poor Risk arm withdrew consent and are not included.
Measure: Number; unit: participants
Arm/Group | Without Grade 3-4 Diarrhea and/or Mucositis | With Grade 3-4 Diarrhea and/or Mucositis
Number analyzed (Participants) | 19 | 16
participants
  CA-CA | 4 | 4
  CA-CC | 7 | 3
  CA-TA | 4 | 4
  CC-CC | 1 | 2
  CC-TA | 2 | 3
  CC-TC | 0 | 0
  TA-TA | 1 | 0

ADVERSE EVENTS:
Time Frame: Beginning of treatment through 30 days after the end of surgery.
Description: Two patients in both the "Good Risk Arm" and the "Poor Risk Arm" withdrew consent and are not included.
Arm/Group | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4)
Serious Adverse Events (participants affected / at risk) | 16/96 | 12/35
Other Adverse Events (participants affected / at risk) | 96/96 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) (N=96) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4) (N=35)
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhea/RT enteritis (Gastrointestinal disorders) | 7 | 7
Perforation/abscess/leak fistula (Gastrointestinal disorders) | 2 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Gastrointestinal bleed (Gastrointestinal disorders) | 1 | 0
Anemia-blood transfusion (Blood and lymphatic system disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hernia repair (Injury, poisoning and procedural complications) | 1 | 0
Crohn's flare (Gastrointestinal disorders) | 1 | 0
Aneurysmal bleed (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Good Risk (Thymidylate Synthase (TYMS)*2/*2, *2/*3, *2/*4) (N=96) | Poor Risk (Thymidylate Synthase (TYMS)*3/*3, *3/*4) (N=35)
Leukocytes (total WBC) (Investigations) | 30 | 20
Platelets (Investigations) | 12 | 1
Hemoglobin (Blood and lymphatic system disorders) | 66 | 30
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 8 | 11
Lymphopenia (Investigations) | 88 | 32
Nausea (Gastrointestinal disorders) | 25 | 19
Vomiting (Gastrointestinal disorders) | 12 | 8
Diarrhea (Gastrointestinal disorders) | 72 | 26
Constipation (Gastrointestinal disorders) | 7 | 6
Dehydration (Metabolism and nutrition disorders) | 6 | 6
Indigestion/cramping (Gastrointestinal disorders) | 13 | 10
Heartburn (Gastrointestinal disorders) | 2 | 1
Tenesmus (Gastrointestinal disorders) | 13 | 1
Rectal spasms (Gastrointestinal disorders) | 1 | 0
Flatus (Gastrointestinal disorders) | 0 | 1
Stomatitis/mucositis (Gastrointestinal disorders) | 34 | 10
Anorexia (Metabolism and nutrition disorders) | 16 | 12
Ileitis/Ileus (Gastrointestinal disorders) | 1 | 1
Bleeding-GI (Gastrointestinal disorders) | 17 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Bilirubin - increased (Investigations) | 26 | 12
SGOT/SGPT - increased (Investigations) | 18 | 13
Alkaline phosphatase - increased (Investigations) | 12 | 7
BUN - increased (Investigations) | 3 | 1
Creatinine -increased (Investigations) | 19 | 6
Dysuria (Renal and urinary disorders) | 14 | 4
Incontinence (Renal and urinary disorders) | 6 | 1
Proteinuria (Renal and urinary disorders) | 3 | 2
Nocturia (Renal and urinary disorders) | 5 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 3
Edema (General disorders) | 3 | 1
Neuropathy - motor (Nervous system disorders) | 0 | 2
Neuropathy-sensory (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 1 | 0
Mood alteration-depression (Psychiatric disorders) | 0 | 2
Mood alteration-anxiety (Psychiatric disorders) | 1 | 2
Seizure (Nervous system disorders) | 0 | 1
Tremors (Nervous system disorders) | 0 | 1
Chills (General disorders) | 3 | 2
Fever without infection (General disorders) | 2 | 3
Sweats (Investigations) | 4 | 0
Fatigue (General disorders) | 27 | 22
Weight loss (Investigations) | 10 | 5
Insomnia (Psychiatric disorders) | 3 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 16 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 13
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 9 | 8
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 13 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 13
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1
Hypoprotenemia (Metabolism and nutrition disorders) | 1 | 0
Skin itching/irritation/rash/desquamation (Skin and subcutaneous tissue disorders) | 50 | 17
Skin dryness (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Flushing (Vascular disorders) | 1 | 0
Erythema/PPE (Skin and subcutaneous tissue disorders) | 20 | 4
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 7 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Infection (Infections and infestations) | 4 | 4
Abscess (Infections and infestations) | 0 | 1
PT (Investigations) | 5 | 2
PTT (Investigations) | 3 | 1
Defibrillator malfunction (Investigations) | 1 | 0
Pain-rectum (Gastrointestinal disorders) | 50 | 24
Pain-head, headache (Nervous system disorders) | 2 | 1
Ocular/vision-eye discomfort (Eye disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes